CLINICAL TRIAL: NCT06169943
Title: A Mhealth Social Support Program on Health Behaviors Among People at Risk of Metabolic Syndrome: a Feasibility Randomized Controlled Trial
Brief Title: Mhealth Social Support for People at Risk of Metabolic Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Lon Tam, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RS-2023-AT
Record Dates: First submitted 2023-12-04; First posted 2023-12-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Syndrome
Keywords: mhealth; metabolic syndrome; lifestyle modifications
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Intervention group Control group
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the participants' group allocation throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Participants in the control group will receive the same mobile app as the intervention group but with limited function.
  Interventions: Other: Control
- Intervention (Experimental): Participants in the intervention group will receive the mHealth social support program.
  Interventions: Other: mHealth social support program

INTERVENTIONS:
Other: mHealth social support program — This is a 3-month program comprises mobile app, group discussion, individual telephone contact, and reminders.
  Arms: Intervention
Other: Control — The same mobile app as the intervention group but with limited function.
  Arms: Control

SUMMARY:
This trial is to examine the feasibility, acceptability, and preliminary effect of a mHealth social support program on lifestyle modifications among people at risk of metabolic syndrome in Hong Kong at 3- and 6-month follow-ups.

DETAILED DESCRIPTION:
Metabolic syndrome is a cluster of unhealthy conditions that affects more than 1 billion people in the world. Lifestyle modifications can reduce the risk to develop metabolic syndrome, while the report showed that over 95% of people in Hong Kong did not practice healthy lifestyle. This trial is to examine the feasibility, acceptability, and preliminary effect of a mHealth social support program on lifestyle modifications among people at risk of metabolic syndrome in Hong Kong. Eighty eligible participants will be recruited from community centers and be randomized into intervention group or control group. Participants in the control group will receive a mobile app with limited function, while those in the intervention group will receive a theory-guided mhealth social support program. Data will be collected at baseline, 3 months, and 6 months on the outcomes of feasibility, acceptability, and lifestyle modifications. Data will be analyzed using a generalized estimating equation based on the intention-to-treat principle. The findings of this study will provide valuable information for a full randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults aged ≥ 45 years
2. With central obesity according to IDF criteria
3. Being treated of hypertension, dyslipidemia, or diabetes
4. Able to give informed consent
5. Attain at least 6 years of formal education
6. Have a smartphone with internet connection and able to use WhatsApp

Exclusion Criteria:

1. Concurrently participating in another clinical trial, lifestyle/dietary intervention, or weight control program
2. Known history of psychiatric disorders

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Physical activity level | Baseline, 3, and 6 months
  Total exercise amount will be quantified with a modified version of the Godin-Shephard Leisure-Time Physical Activity Questionnaire.

SECONDARY OUTCOMES:
Healthy eating | Baseline, 3, and 6 months
  Diet subscale of the Chinese version of Health Promoting Lifestyle Profile II. The subscale includes eight items measuring healthy eating on a 4-point Likert scale (1=never to 4=routinely), ranged from 8-32. The higher sum score indicates more adoption of healthy eating.
Metabolic syndrome knowledge | Baseline, 3, and 6 months
  Chinese version of metabolic syndrome knowledge scale. 10 items cover three domains: definition and diagnosis (5 items), complications (2 items), and preventions (3 items); a higher sum score indicates better understanding of metabolic syndrome.
Perceived social support | Baseline, 3, and 6 months
  Chinese version of multidimensional scale of perceived social support. 12 items measuring perceived support from family and friends; 7-point Likert scale (1=strongly disagree to 7=strongly agree), ranged from 12 -84; a higher sum score indicates more social support is perceived.
Self-efficacy | Baseline, 3, and 6 months
  Nutrition and Exercise subscale of the Chinese version of Self-rated Abilities for Health Practices.
  7 items measuring diet self-efficacy and 7 items measuring PA self-efficacy; five-point Likert scale (0=not confident to 4=very confident) that a higher score indicates higher confidence to adopt lifestyle modifications in daily life.
Blood pressure | Baseline, 3, and 6 months
  Both systolic blood pressure and diastolic blood pressure will be measured by a validated and reliable upper-arm automated system (in mmHg) after resting for 20 minutes; an average of two measurements with 1-minute apart is recorded.
Waist circumference | Baseline, 3, and 6 months
  Measured in the nearest 0.1 centimeter.
Body weight | Baseline, 3, and 6 months
  Measured in the nearest 0.1 kilogram.
Body fat mass percentage | Baseline, 3, and 6 months
  Body fat mass percentage will be assessed by a calibrated digital body composition monitor.

IPD SHARING:
Plan to Share IPD: No